CLINICAL TRIAL: NCT04116476
Title: An Open-label, Single-center, Parallel-group Study to Assess Pharmacokinetics, Safety, and Tolerability of a Single Dose of MT-7117 in Subjects With Normal and Impaired Hepatic Function
Brief Title: Study to Assess Pharmacokinetics, Safety, and Tolerability of MT-7117 in Subjects With Normal and Impaired Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanabe Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MT-7117-A02
Record Dates: First submitted 2019-10-03; First posted 2019-10-04 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Mild and Moderate Hepatic Impairment
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Moderate Hepatic Impairment (Experimental)
  Interventions: Drug: MT-7117
- Normal Healthy Matches (Experimental)
  Interventions: Drug: MT-7117
- Mild Hepatic Impairment (Experimental)
  Interventions: Drug: MT-7117

INTERVENTIONS:
Drug: MT-7117 — Single Dose of MT-7117

SUMMARY:
An Open-label, Single-center, Parallel-group Study to Assess Pharmacokinetics, Safety, and Tolerability of a Single Dose of MT-7117 in Subjects with Normal and Impaired Hepatic Function

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 18 to 75 years of age inclusive
* BMI 18 -35 kg/m2
* If female, you are nonpregnant, non-lactating and willing to utilize approved methods of birth control.

Exclusion Criteria:

* Subjects who have mild or moderate hepatic impairment according to Child-Pugh classification system at Screening (except normal healthy matches)
* Subjects who have a known clinically significant (CS) hypersensitivity to MT-7117 or related compounds, including melatonin.
* Subjects who have previously participated in a study involving MT-7117 or taken any other investigational drug within 30 days or 5 half-lives prior to the first dose of IMP, whichever is longer.
* Subjects who have a CS or unstable neurological, renal, cardiovascular, gastrointestinal, pulmonary, or hematologic disease for 14 days prior to enrollment.
* Subjects who have used any prescription or over-the-counter (OTC) medication within 14 days prior to first dose of IMP, except for occasional use of acetaminophen (< 1 g/day for normal hepatic subjects, and < 2 g/day for hepatically impaired subjects) or any other medication approved by the sponsor (a case-by-case basis). For hepatic impaired subjects, prescribed medication or OTC may be permitted by the Investigator and sponsor on a case-by-case basis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-02-16 (Actual); Study Completion 2021-02-16 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of MT-7117 | 0-96 Hours
Area under the plasma concentration time curve from time zero to the time of last quantifiable concentration (AUC0-last) of MT-7117 | 0-96 Hours
Area under the plasma concentration time curve from time zero to infinity (AUC0-∞) of MT-7117 | 0-96 Hours

SECONDARY OUTCOMES:
Time to reach maximum plasma concentration (tmax) of MT-7117 | 0-96 Hours
Plasma terminal elimination half-life (t1/2) of MT-7117 | 0-96 Hours
Apparent oral clearance (CL/F) of MT-7117 | 0-96 Hours
Apparent volume of distribution (Vz/F) of MT-7117 | 0-96 Hours
fraction of unbound drug in plasma or serum (fu) of MT-7117 | 0-96 Hours
Number of participants with Adverse events (AEs) and Serious Adverse Events (SAEs) | 0-96 Hours

CONTACTS AND LOCATIONS:
Overall Officials: Head of Medical Science, Study Director — Tanabe Pharma America, Inc.
Locations (1):
- University of Miami Clinical Pharmacology Unit, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ogasawara A, Ide R, Inoue S, Teng R, Kawaguchi A. Effect of Hepatic and Renal Impairment on the Pharmacokinetics of Dersimelagon (MT-7117), an Oral Melanocortin-1 Receptor Agonist. Clin Pharmacol Drug Dev. 2024 Jul;13(7):729-738. doi: 10.1002/cpdd.1413. Epub 2024 May 15. PMID 38746989